CLINICAL TRIAL: NCT05193760
Title: Robustness Check of Placement and Measurement Algorithms for Blood Flow Measurement on Common Carotid Artery
Acronym: RAdiUS
Status: Completed | Type: Observational
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Collaborators: Philips Electronics Nederland BV (Industry)
Responsible Party: Principal Investigator, Esmée de Boer, Doctoral Candidate, Catharina Ziekenhuis Eindhoven
Other Study IDs: ICBE 2-35542; nWMO-2021.081 (Other: MEC-U)
Record Dates: First submitted 2021-12-23; First posted 2022-01-18 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease; Aortic Valve Disease; Mitral Valve Disease
Keywords: Common carotid artery; Ultrasound
MeSH Terms: conditions — Coronary Artery Disease; Aortic Valve Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is set up to test the robustness of algorithms and models and to optimize them. Furthermore, data are used to investigate the influence of probe orientation on parameters of the common carotid artery.

DETAILED DESCRIPTION:
This study has four objectives:

1. Determine the robustness of the placement and measurement algorithms with ultrasound images, obtained with different ultrasound system settings and probe movements.
2. Verificate and optimize the arterial blood flow model.
3. Determine the variation in location and size of the arteries and veins in the area around the common carotid artery.
4. Determine the influence of probe orientation on parameters obtained from ultrasound measurements of the common carotid artery.

Sample size and missing data Due to limited time in the operating room, the measurement protocol is divided into four parts. Per protocol part data of 25 patients is deemed sufficient to be able to answer the above-mentioned objectives, which would result in a total of 100 inclusions. However, the investigators expect to perform more than one measurement protocol per patient, due to which a total of 75 inclusions is needed. Patients of whom the data is qualitatively too low to be used for analysis will be replaced. As such, the investigators make sure to have qualitatively good data of 25 patients per protocol part.

ELIGIBILITY:
Inclusion Criteria:

* Adult (>18 years) patients.
* Participant should be able to provide informed consent in Dutch.

Exclusion Criteria:

* Participant has a known stenosis of the carotid artery.
* Patient has open wounds in the measurement area (area in the neck around the carotid artery).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (>18 years) cardiac surgery or TAVI patients.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
Robustness of placement and measurement algorithms. | During data acquisition, which is pre-surgery.
  Using the obtained US images of the common carotid artery, the robustness of our algorithms for placement and measurements will be checked.
Verify and improve the arterial blood flow model. | During data acquisition, which is pre-surgery.
  Using the obtained US images of the common carotid artery, our arterial blood flow model will be verified and adapted.
Orientation of ultrasound probe. | During data acquisition, which is pre-surgery.
  Using the obtained US images of the common carotid artery, the influence of probe orientation on carotid artery parameters will be investigated.

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Bouwman, MD PhD, Principal Investigator — Catharina Ziekenhuis Eindhoven; John van Rooij, MSc, Study Chair — Philips Electronics Nederland B.V.
Locations (1):
- Catharina Ziekenhuis Eindhoven, Eindhoven, North Brabant, Netherlands